CLINICAL TRIAL: NCT03045211
Title: Post-Physical Therapy Extension of In-Home Dynamic Standing Table Use in Parkinson Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Michigan (Other)
Responsible Party: Principal Investigator, Nicolaas Bohnen, MD, PhD, Professor, University of Michigan
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: HUM00118467
Record Dates: First submitted 2017-01-31; First posted 2017-02-07 (Estimated); Last update posted 2020-09-22 (Actual); Status verified 2020-09

CONDITIONS: Parkinson Disease
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- In-Home Standing Table (Experimental): Participants in this arm will receive a dynamic standing table to be used in their home for at least two hours per day for at least five days per week for a 16-week period. Specific activities will be tracked with a logbook. PD subjects will be coached by a physical therapist on proper body positioning at the table, use of anti-fatigue mat, and optimal monitor height. The physical therapist will adhere to the "neutral body positioning" guidelines as provided by the OSHA. The physical therapist will also perform an in-home safety assessment of the office or room in which the table will be placed to ensure safety not only for the users but also for family members or children. The physical therapist will monitor each participant throughout the study by making biweekly compliance phone calls.
  In addition, this group will received standard of care, which is weekly group exercise sessions during the 16-week period of table use.
  Interventions: Device: Dynamic Standing Table
- Standard of Care (No Intervention): this group will received standard of care only, which is weekly group exercise sessions during a 16-week period. Instructions, coaching, and compliance phone calls will also be provided to the participants of this arm such that both arms have the same amount of contact time with the physical therapist.

INTERVENTIONS:
Device: Dynamic Standing Table — The dynamic standing table is a height-adjustable standing table which gives periodic cues to the user to make stepping movements.
  Arms: In-Home Standing Table

SUMMARY:
When postural imbalance and gait difficulties emerge in subjects with Parkinson disease, patients are typically referred for a number of physical therapy sessions. However, there is a critical gap in clinical practice on what to do once patients have completed their therapy sessions. To fill this gap, the study team has developed a standing table with a tabletop system that encourages weight shifting during upright standing ("dynamic standing table"), and therefore may be a unique means to increase daily physical activity by integrating the system with routine desktop activities of daily living. The purpose of this study is to determine whether a post-physical therapy in-home physical activity program using the dynamic standing table (as an adjunct to post-physical therapy standard of care-weekly physical activity group sessions) is effective in sustaining the mobility benefits of physical therapy in individuals with Parkinson disease.

DETAILED DESCRIPTION:
Axial motor dysfunctions in Parkinson disease (PD) are least responsive to dopaminergic therapy and incline many patients towards a sedentary lifestyle. This places PD patients at increased risk for the negative consequences of physical inactivity. When PD patients develop postural imbalance and gait difficulties, including falls, they are generally referred to physical therapy for optimal management. Although these patients do benefit from physical therapy, there is a critical gap in clinical practice on what to do next once the physical therapy sessions are over. Clinical experience shows that most patients return to a sedentary lifestyle indicating an urgent need for post-physical therapy in-home physical activity programs in PD with postural imbalance and gait difficulties to preserve mobility functions. Recent advances in physical activity research tout non-exercise physical activity approaches to promote healthy lifestyle modifications. Non-exercise physical activities are activities of daily living, like cleaning, shopping, and standing, other than intentional exercise. For PD patients with postural imbalance and gait difficulties, normal upright standing and weight-shifting (stepping) for longer periods of time may be an ideal form of non-exercise physical activity. It activates lower extremity muscles and encourages postural activity. To promote this type of non-exercise physical activity, the study team applies a "dynamic standing table", which periodically cues users to make steps. Dynamic standing would represent a minimal level of physical activity compared to sitting, which is pervasive in PD subjects with postural imbalance and gait difficulties. Use of the dynamic standing table can easily be incorporated with routine desktop activities, such as computer use, reading, or watching TV and may promote physical activity. The purpose of this study is to determine whether a post-physical therapy in-home physical activity program using the dynamic standing table (as an adjunct to post-physical therapy standard of care-weekly physical activity group sessions) is effective in sustaining the mobility benefits of physical therapy compared with post-physical activity standard of care alone in individuals with Parkinson disease and postural imbalance and gait difficulties. The study team is testing the exploratory hypothesis that post-physical therapy gains in mobility functions in PD patients with postural imbalance and gait difficulties will be preserved better with in-home dynamic standing table use compared to a control group. After consulting with regulatory specialists, this device was determined to be 510k exempt and falls under part 890 Physical Medicine devices Subpart F- Physical Medicine therapeutic devices. Sec. 890.5370 Nonmeasuring exercise equipment.

ELIGIBILITY:
Inclusion Criteria:

* Presence of Parkinson's disease. PD diagnosis following the UK Parkinson's Disease Society Brain Bank Research Center (UKPDSBRC) clinical diagnostic criteria for PD, consistent with the typical nigrostriatal denervation pattern on VMAT2.
* Hoehn and Yahr stages 2-4 and/or presence of PIGD features, such as history of (near) falls, slow gait, and/or freezing of gait.
* Available space to place table in their home (approximately 6 ft x 5 ft area).

Exclusion Criteria:

* Inability to stand or walk without an assistive device.
* History of symptoms in stance that preclude safe and comfortable participation, such as dizziness and lightheadedness, orthostasis, severe symptomatic leg or back musculoskeletal pain.
* History of significant symptomatic cardiovascular or pulmonary disease.
* History of active symptomatic rheumatic arthritis.
* History of stroke or other focal brain conditions with residual sensorimotor deficits interfering with stance functions.
* History of chronic pain syndrome requiring daily narcotic analgesics.
* Evidence of dementia.
* Venous stasis or severe varicosities

Min Age: 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2016-09 (Actual); Primary Completion 2020-03 (Actual); Study Completion 2020-04 (Actual)

PRIMARY OUTCOMES:
Change in stride velocity during the instrumented Timed Up and Go test from week 6 to week 23 | At week 6 (post-physical therapy); at week 23 (post 16-week table intervention)
  Instrumented Timed Up and Go, Subject starts in seated position rises from chair and walks 3 meters, then returns to chair in a seated position

CONTACTS AND LOCATIONS:
Overall Officials: Nicolaas Bohnen, MD PhD, Principal Investigator — University of Michigan
Locations (1):
- University of Michigan Functional Neuroimaging, Cognitive and Mobility Laboratory, Ann Arbor, Michigan, United States

IPD SHARING:
Plan to Share IPD: No